CLINICAL TRIAL: NCT06844838
Title: FASt Track in Elective Neurosurgery: the Role of Low Propofol Bis-NOL Guided General Anaesthesia for Full, Early and Safe Awakening
Acronym: FasTrack
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: FasTrack
Record Dates: First submitted 2025-02-07; First posted 2025-02-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Supratentorial Brain Tumor Surgery
Keywords: General Anaesthesia; BIS; Bispectral Index; NOL; Nocipection Level; Neuroanesthesia; Target Colled Infusion TCI; Craniectomy; Awakening; ERAS; Fast Track; Propofol; Remifentanil; Pain; Nociception; RASS
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the effect of intraoperative sedation dosage on awakening and recovery of consciousness after elective neurosurgical surgery.

DETAILED DESCRIPTION:
The project will have a total duration of 24 months and will mainly consist of a data collection phase (months 1-24) and a data analysis and results publication phase (months 15-24). Preoperative clinical and socio-demographic data will be collected from patients' medical records. Psychological variables will be administered to the patient before elective neurosurgical surgery.

BIS-guided general anesthesia will be induced by administering sedative and analgesic drugs to the effector site Ce (Effect Site) by target-controlled infusion (TCI). Propofol and remifentanil will be titrated to maintain blood pressure, body temperature, pCO2 and SaO2 in a normal range and BIS values between 40 and 60. Pharmacological data will be relevant at the end of the intervention from the drug infusion pumps. The Recovery Room multidisciplinary team will assess the quality of awakening following the Awakening Chart (Figure 1). This assessment involves dichotomous scoring (yes/no; correct/incorrect) of specific items. To assess the recovery of consciousness, during the pre-extubation phase, simple requests/questions will be asked of the patient: show tongue; show two fingers; give phone number; state place; identify what day is today; report date of birth; notify residence; perform simple multiplication (e.g., 4x5). The following variables will be collected during the periestubation phase: cough, blood pressure ± 20% of baseline, chills, NRS > 3, RASS < -1 or > 0. An abbreviated version of the STAI questionnaire will also be administered to the patient to assess anxiety on awakening. Awakening is considered good and optimal only if a score of 13 is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients with supra- and sub tentorial neurosurgical pathology who meet the following inclusion criteria will be enrolled:
* Age greater than or equal to 18 years

Exclusion Criteria:

* Psychiatric illness in history and/or taking psychotropic drugs
* Glasgow Coma Score (GCS) < 15
* Presence of overt cognitive decline or speech disorders
* Patients younger than 18 years of age
* Intraoperative hypothermia (< 36°)
* Intraoperative hypotension (MAP < 20% of baseline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing neurosurgical surgery afferent to the Department of Neurosurgery of the IRCCS Carlo Besta Neurological Institute Foundation will be consecutively enrolled from the date of study approval for 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
General Anaesthesia effect on Awakening | 2 years
  Correlation between intraoperative dosage of Propofol and Remifentanil with respect to dichotomous outcome related to quality of awakening post GA.

SECONDARY OUTCOMES:
RASS Scale score | 2 years
  RASS (Richmond Assesmenet sedation scale) scale score at post-GA awakening Analysis of the association between perioperative indicators - age, BMI, Milan Complexity Score, APAIS - and outcome on awakening. The minimum RASS scale is - 5 (unresponsive patient after painfull stimulation) and the maximum is + 4 (comactive patient). The optimal RASS scale is 0/-1.
NRS scale score | 2 years
  NRS (Numerical rating scale ) scale score at post-GA awakening Analysis of the association between perioperative indicators - age, BMI, Milan Complexity Score, APAIS - and outcome on awakening. The minimum NRS scale is 0 (no pain at all) and the maximum is 10 (the maximum pain ever suffered)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No